CLINICAL TRIAL: NCT00725205
Title: Patient Compliance During PegIntron (Injection Pen) and Rebetol Combination Therapy in Chronic Hepatitis C
Brief Title: Patient Compliance During PegIntron and Rebetol Combination Therapy in Chronic Hepatitis C (Study P04690)
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: P04690
Record Dates: First submitted 2008-07-25; First posted 2008-07-30 (Estimated); Results first posted 2011-11-18 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-10

CONDITIONS: Hepatitis C, Chronic; Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chronic hepatitis C participants: Untreated chronic hepatitis C (CHC) participants starting Peginterferon alfa-2b (injection pen) and Ribavirin combination therapy as their usual medical treatment according to the approved dosage/regimen were selected for this study.
  Interventions: Biological: PegIntron (Peginterferon alfa-2b); Drug: Rebetol (Ribavirin)

INTERVENTIONS:
Biological: PegIntron (Peginterferon alfa-2b) — Peginterferon alfa-2b (injection pen) administered according to the product's labeling and current practice in Hungary (1.5 micrograms [mcg]/killogram [kg]) for 12 weeks. Those participants whose continued treatment was warranted beyond week 12 based on response received therapy for 24 or 48 weeks depending on the viral genotype.
  Other Names: PegIntron; SCH 54031
Drug: Rebetol (Ribavirin) — Ribavirin capsules administered according to the product's labeling and current practice in Hungary (weight based daily) for 12 weeks. Those participants whose continued treatment was warranted beyond week 12 based on response received therapy for 24 or 48 weeks depending on the viral genotype.
  Other Names: Rebetol; SCH 18908

SUMMARY:
Participants will receive PegIntron injection pen (Peginterferon alfa-2b) and Rebetol (Ribavirin) combination therapy as their usual medical treatment. The current study aims to evaluate whether the previously introduced, and now widely accepted and implemented educational program, which represents additional efforts in everyday practice to increase patient compliance, will succeed in achieving adherence rate in treated participants similar to the extent demonstrated by clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Before inclusion, all participants must be informed and must give consent for the use of his/her anonymized health data related to his/her treatment with Peginterferon alfa-2b (injection pen) and Ribavirin.

Exclusion Criteria:

* According to Peginterferon alfa-2b/Ribavirin label.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Untreated chronic hepatitis C (CHC) participants starting Peginterferon alfa-2b (injection pen) and Ribavirin combination therapy as their usual medical treatment according to the approved dosage/regimen were selected for this study.
Sampling Method: Non-Probability Sample
Enrollment: 294 (Actual)
Dates: Start 2006-03; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 294 participants were enrolled, 2 participants were not treated.
Groups:
- Peginterferon Alfa-2b and Ribavirin: Previously untreated Chronic Hepatitis C (CHC) participants treated with a treatment regimen of 1.5 micgrograms (mcg)/killogram (kg) Peginterferon alfa-2b (injection pen) and weight based daily Ribavirin capsules combination therapy as their usual medical treatment administered according to the product's labeling and current practice in Hungary for 12 weeks. Those participants whose continued treatment was warranted beyond Week 12 based on response received therapy for 24 or 48 weeks depending on the viral genotype.
Period: Overall Study
Arm/Group | Peginterferon Alfa-2b and Ribavirin
Started | 294
Completed | 207
Not Completed | 87
Not completed — Adverse Event | 22
Not completed — Investigator Discontinued | 1
Not completed — Non-compliance With Protocol | 14
Not completed — Other | 8
Not completed — Protocol Defined Clinical Event | 1
Not completed — Treatment Failure | 41

BASELINE CHARACTERISTICS:
Groups:
- Peginterferon Alfa-2b and Ribavirin: Previously untreated CHC participants treated with a treatment regimen of 1.5 mcg/kg Peginterferon alfa-2b (injection pen) and weight based daily Ribavirin capsules combination therapy as their usual medical treatment administered according to the product's labeling and current practice in Hungary for 12 weeks. Those participants whose continued treatment was warranted beyond Week 12 based on response received therapy for 24 or 48 weeks depending on the viral genotype.
Arm/Group | Peginterferon Alfa-2b and Ribavirin
Number analyzed (Participants) | 294
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.7 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 165
  Male | 129

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Are Triple-80 Compliant
Description: Participants who continued treatment beyond Week 12 (i.e., 24 or 48 weeks depending on the viral genotype) were assessed for triple-80 compliance. Triple-80 compliant, or simply compliant, participants were those that received >= 80% of the planned total doses of both pegylated interferon alfa-2b and ribavirin for >=80% of the duration of the therapy. 3 rates were computed: Compliance with study duration, compliance with pegylated interferon dose, and compliance with ribavirin dose. A participant was defined as triple-80 compliant, if none of the 3 rates as defined above were less than 80.
Time Frame: 24 or 48 Weeks
Population: All enrolled participants who received any dose of any medication, had a known viral genotype, and did not discontinue from the study with the status being "treatment
  failure". Of the 294 enrolled participants, 253 participants started treatment and continued treatment beyond Week 12.
Measure: Number; unit: Participants
Arm/Group | Peginterferon Alfa-2b and Ribavirin
Number analyzed (Participants) | 253
Participants | 183

2. Secondary Outcome: Number of Participants Who Achieved Sustained Virological Response as Assessed at 24-week Post-treatment Follow-up
Description: Sustained virologic response (SVR) was assessed at post-treatment Follow-up Week 24. Day 1 of the Follow-up period was defined as the first day after the last dose day. A participant was considered a sustained responder if the participant had undetectable Hepatitis C virus Ribonucleic acid (HCV-RNA) level (based on qualitative test result) at Follow-up Week 24. If a participant with missing polymerase chain reaction (PCR) data at Follow-up Week 24 had undetectable HCV-RNA level at Follow-up Week 12, the participant was also considered as a sustained responder.
Time Frame: 24 Weeks following completion of 24 or 48 weeks of therapy
Population: Full Analyses Set: All enrolled participants who received any dose of any medication (Peginterferon or Ribavirin) and had a known viral genotype. Of the 294 enrolled participants, 2 were not treated.
Measure: Number; unit: Participants
Arm/Group | Peginterferon Alfa-2b and Ribavirin
Number analyzed (Participants) | 292
Participants | 66

3. Secondary Outcome: Number Of Participants Self-Administering Pegylated Interferon Alfa-2b
Description: Number of participants self-administering Pegylated interferon alfa-2b injection pen. If a participant changed the way he or she administered the injection pen during the course of the study (from self-administering to clinic-administering or the other way around), that participant was also considered as self-administering.
Time Frame: Up to 48 Weeks
Population: All Participants enrolled.
Measure: Number; unit: Participants
Arm/Group | Peginterferon Alfa-2b and Ribavirin
Number analyzed (Participants) | 294
Participants | 291

ADVERSE EVENTS:
Description: The All Patients as Treated (APAT) population included all enrolled participants who took at least one dose of Peginterferon alfa-2b or Ribavirin.
Arm/Group | Peginterferon Alfa-2b and Ribavirin
Serious Adverse Events (participants affected / at risk) | 9/292
Other Adverse Events (participants affected / at risk) | 109/292
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Peginterferon Alfa-2b and Ribavirin (N=292)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Eosinophilia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Hepatic Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Depression (Psychiatric disorders) | 1 (1)
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Toxic Skin Eruption (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Peginterferon Alfa-2b and Ribavirin (N=292)
Anaemia (Blood and lymphatic system disorders) | 74 (87)
Thrombocytopenia (Blood and lymphatic system disorders) | 15 (17)
Pyrexia (General disorders) | 23 (26)
Weight Decreased (Investigations) | 19 (19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators require the SPONSOR'S written permission to publish any information pertaining to the study during and five years after closure of the study.